CLINICAL TRIAL: NCT00827424
Title: The Impact of the PACE Program Implementation on Health Services Utilization by Obese Arab Women (The AWESOME Study: Arab WomEn Study on Obesity Metabolism and Exercise)
Brief Title: The Impact of the PACE Program Implementation on Health Services Utilization by Obese Arab Women
Acronym: AWESOME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clalit Health Services (Other)
Responsible Party: Batya Kornboim MD, Clinical Research Unit, Clalit Health Services, Haifa and Western Galilee District
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMC-07-0054CTIL
Record Dates: First submitted 2009-01-21; First posted 2009-01-22 (Estimated); Last update posted 2010-08-24 (Estimated); Status verified 2010-08

CONDITIONS: Obesity
Keywords: physical activity (PA); obesity; life style modification; physical activity; diet; BMI reduction; clinical and metabolic measure; health expenditure; improvement of patient readiness for lifestyle change
MeSH Terms: conditions — Obesity; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): This arm will receive Lifestyle counseling by applying a modified PACE protocol
  Interventions: Behavioral: Lifestyle counseling by applying a modified PACE protocol
- 2 (No Intervention): Subject in this arm will be recruited but will receive no intervention

INTERVENTIONS:
Behavioral: Lifestyle counseling by applying a modified PACE protocol — Lifestyle counseling by applying a modified PACE protocol to obese Arab women
  Arms: 1

SUMMARY:
Scientific background:

Obesity is a known risk factor for cardiovascular disease, metabolic syndrome, and diabetes. In Israel, the prevalence of obesity and diabetes among Arab females is 2 and 2.8 times higher than Jewish females, respectively. The economic impact of obesity and overweight in terms of illness, disease and lost productivity is estimated to amount to 2-9% of the national health budget in countries with high GDP. Diabetics have medical expenditure that is 2.4 times higher than non diabetics per capita.

Lifestyle modification is an effective tool in reducing morbidity and health care expenditure but despite that most family practitioners usually treat the complications of obesity rather than preventing it.

PACE is a comprehensive health promotion guide in counseling patients to an active healthy lifestyle. PACE is designed to assist the primary health care providers to promote physical activity and dietary changes during routine office visits.

Objectives:

To asses the impact of PACE program on increasing the amount of physical activity, improving clinical and metabolic indices, increasing the documentation of lifestyle indices in the medical records and reducing health care expenditure and utilization.

Working hypothesis:

Implementing a modified PACE protocol can achieve this objectives in Arab women.

Methodology:

The investigators will conduct a structured, multidisciplinary and continuous primary care based intervention, assisted by trained health promoters and applying a locally adjusted PACE protocol.

ELIGIBILITY:
Inclusion Criteria:

* Arab women
* Age range 35-64
* Insured by Clalit Health Services (CHS)
* Residence in the target communities
* BMI > 30 kg/m2
* Signed informed consent

Exclusion Criteria:

* Failure in any of the inclusion criteria

Ages: 35 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2008-12; Primary Completion 2010-05 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
A significant change in BMI | every 3 months for 18 month

SECONDARY OUTCOMES:
Patient's lifestyle habits: physical activity, eating habits | every 3 months for 18 month
Patient's clinical measures: BP, Waist Circumference | every 3 months for 18 month
Patient's metabolic measure: HbA1c, lipid profile, fasting plasma glucose (FPG) | every 3 months for 18 month
Patient's readiness for change: Determined by the PACE score | every 3 months for 18 month

CONTACTS AND LOCATIONS:
Overall Officials: Batya Kornboim, MD, Principal Investigator — Clinical Research Unit, Clalit Health Services, Haifa and Western Galilee District .; Uzi Milman, MD, Principal Investigator — Clinical Research Unit, Clalit Health Services, Haifa and Western Galilee District .
Locations (1):
- Clinical Research Unit, Clalit Health Services, Haifa and Western Galilee District ., Haifa, Israel